CLINICAL TRIAL: NCT02713334
Title: Cancer Patients Decision Making and Family Communication About Secondary Findings From Tumor Genomic Profiling
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-080
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Tumor Genomic Profiling
Keywords: Decision Making; Communication; 16-080
MeSH Terms: conditions — Communication | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: survey
Behavioral: semi-structured interview

SUMMARY:
The objective of this protocol is to characterize cancer patients' responses to learning their secondary findings arising from tumor genomic profiling, and the process and outcomes of their decisions to communicate these results to their families.

DETAILED DESCRIPTION:
For Phase 1 of this study, the investigators will conduct a prospective, observational study with cancer patients undergoing tumor genomic profiling (n = 300) and their family members (anticipated n ≈ 150). Data collection will occur through an embedded mixed methods design, in which both quantitative (i.e., survey) and qualitative (i.e., semi-structured interview) data are collected at the same timepoint in order to obtain a more complete understanding of specific processes and outcomes.

They will be recruited from those who already enrolled in protocol #12-245, and who agree to receive their secondary findings through Consent Part C of this existing protocol.

For Phase 2 of this study, participants (n=500) who have received pathogenic secondary findings through protocol #12-245 will be recruited.

For Phase 3, efforts will be expanded from the adult populations explored in the preceding phases to the experiences of patients affected by pediatric cancers and their families. Cross-sectional mixed methods data from AYA survivors of pediatric cancers (n=50) and adult caregivers of survivors of pediatric cancer (n=50) will be collected.

ELIGIBILITY:
Inclusion Criteria:

Patients (Phase I):

* 18 years of age or older
* Has consented to MSK IRB protocol #12-245, Consent A and Part C
* Has not received secondary findings as a result of MSK IRB protocol #12-245, Consent Part C as per EMR and/or patient report
* Diagnosed with a solid tumor as per EMR and/or clinician judgment
* English-fluent; the surveys were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the surveys.

Family members (Phase I):

* 18 years of age or older as per self report
* Nominated by the patient participant as a family member with whom the secondary findings have been shared (spouses/partners are eligible as "family members" for the purposes of this study)
* English-fluent; the surveys were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the surveys.

Patients (Phase 2):

* 18 years of age of older
* Has consented to MSK IRB protocol #12-245, Consent Part A and C
* English-fluent; the surveys were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefor, participants must be able to communicate in English to complete the surveys.

AYA Survivors of Pediatric Cancers (Phase 3):

* Age 15 to 30 years old
* Are at least 1 year post-treatment for pediatric cancer (i.e., any cancer diagnosed before age 18)
* Has consented or provided assent to MSK IRB protocol #12-245, Consent Part A and C
* Has received pathogenic secondary findings as a result of MSK IRB protocol #12- 245, Consent Part C as per EMR and/or CGS care provider report
* Participated in a CGS consultation following receipt of secondary findings
* English-fluent; the surveys were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the surveys.

Adult Caregivers of Survivors of Pediatric Cancers (Phase 3):

* 18 years of age or older
* Are the caregiver of a child who was treated for pediatric cancer (i.e., any cancer diagnosed before age 18). Caregiver status is based on either: 1) nomination as such by a young adult survivor (i.e., age 18+), 2) having consented on behalf of a minor child (i.e., age <18) to MSK IRB protocol

  #12-245 Part A and C plus self-reported confirmation that s/he is the caregiver for the child, or 3) nomination by the adult who consented on behalf of a minor child (i.e., age <18) to MSK IRB protocol #12-245 Part A and C plus self-reported confirmation that s/he is the caregiver for the child
* That child is currently alive and at least 1 year post-treatment for pediatric cancer (i.e., any cancer diagnosed before age 18)
* Has consented on behalf of that child, or that child consented, to MSK IRB protocol #12-245, Consent Part A and C
* That child received pathogenic secondary findings as a result of MSK IRB protocol #12-245, Consent Part C as per EMR and/or CGS healthcare provider report
* Participated in a CGS consultation following receipt of secondary findings
* English-fluent; the surveys were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the surveys

Exclusion Criteria:

* Received genetic testing in the past that resulted in a pathogenic finding or a variant of unknown significance as reported in the EMR.
* Major psychiatric illness or cognitive impairment that in the judgment of the investigator or study staff would preclude study participation
* Any patients who are unable to comply with the study procedures as determined by the study investigators or study staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 300 participants for the proposed study from those already enrolled in protocol #12-245, and who agree to receive their secondary findings through Consent Part C of this existing protocol.
Sampling Method: Non-Probability Sample
Enrollment: 495 (Actual)
Dates: Start 2016-02-25; Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
The investigators will assess patients' emotional responses to receiving their secondary findings | 1 year
  Through quantitative (i.e., survey) assessments, the investigators will assess patients' emotional (both positive and negative) responses to receiving their secondary findings, and their perceptions regarding the utility of this information and communicating it to family.

CONTACTS AND LOCATIONS:
Overall Officials: Jada Hamiliton, PhD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/